CLINICAL TRIAL: NCT06949566
Title: Evaluation of Grip Strength and Reaction Time Following Induced Fatigue of the Wrist Flexors: The Acute Effects of Local Vibration
Brief Title: Post-Fatigue Vibration: Impact on Grip and Reaction Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Omer Dursun, Asst. Prof., Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BEUFTR-8
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Muscle Fatigue
Keywords: Local Vibration; Upper Extremity Function; Wrist Flexors; Neuromuscular Performance

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The evaluator and the researcher administering the plantar vibration intervention will be different. Patients will be blinded to their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham Vibration Group (Sham Comparator): In this group, sham vibration will be administered following the muscle fatigue protocol. The vibration device will be activated but positioned close to the muscle without direct contact for a duration of 10 minutes. Participants will be told that they are receiving treatment with an electromagnetic vibration device.
  Interventions: Other: Sham Local Vibration
- 50 Hz Local Vibration Intervention Group (Experimental): Participants in this group will receive 50 Hz local vibration following the muscle fatigue protocol. The local vibration will be applied along the flexor carpi ulnaris muscle for a duration of 10 minutes.
  Interventions: Other: 50 Hz Local Vibration
- 100 Hz Local Vibration Intervention Group (Experimental): Participants in this group will receive 100 Hz local vibration following the muscle fatigue protocol. The local vibration will be applied along the flexor carpi ulnaris muscle for a duration of 10 minutes.
  Interventions: Other: 100 Hz Local Vibration

INTERVENTIONS:
Other: 100 Hz Local Vibration — Participants in this group will receive 100 Hz local vibration along the flexor carpi ulnaris muscle for a duration of 10 minutes.
  Arms: 100 Hz Local Vibration Intervention Group
Other: 50 Hz Local Vibration — Participants in this group will receive 50 Hz local vibration along the flexor carpi ulnaris muscle for a duration of 10 minutes.
  Arms: 50 Hz Local Vibration Intervention Group
Other: Sham Local Vibration — Participants in this group will receive sham vibration following the muscle fatigue protocol. The vibration device will be turned on but held near the muscle without making contact for 10 minutes. Participants will be informed that they are being treated with an electromagnetic vibration device.
  Arms: Sham Vibration Group

SUMMARY:
This study aims to investigate the acute effects of local vibration applied after induced fatigue of the wrist flexor muscles on grip strength and upper extremity reaction time.

DETAILED DESCRIPTION:
This randomized controlled study will be conducted with a minimum of 42 participants who meet the inclusion and exclusion criteria. Participants will be randomly assigned to one of three groups: control, 50 Hz local vibration, or 100 Hz local vibration.

ELIGIBILITY:
Inclusion Criteria:

1. Female individuals aged 18-25

Exclusion Criteria:

1. Having an open wound in the area where local vibration is applied
2. A history of previous or current upper extremity injury
3. Use of anti-inflammatory drugs
4. Having a diagnosis of epilepsy

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Individuals who self-identify as female.
Enrollment: 42 (Actual)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Hand Grip Strength Measurement | Change in hand grip strength from baseline following intervention or rest
  Grip strength will be assessed using a JAMAR® hydraulic hand dynamometer, which has five grip positions. The test will follow American Society of Hand Therapists guidelines, with the elbow at 90° flexion.
  Measurements will be taken on the dominant hand. Participants will sit with their head facing forward, shoulders slightly abducted (10-20°), elbows at 90°, and wrists and hands in a neutral position. Both upper extremities will remain relaxed, and feet will be flat on the floor.
  Fingers will be fully extended and adducted. Participants will be instructed not to allow their hands or forearms to touch the body. The dynamometer will be adjusted to fit the participant's hand size, typically set at the second handle position.
Upper Extremity Reaction Time Measurement | Change in upper extremity reaction time from baseline following following intervention or rest
  Upper extremity reaction times will be recorded using the BlazePod system (Play Coyotta Ltd., Tel Aviv, Israel). Participants will begin the reaction time test while seated, with both hands placed on a table, palms facing downward, and elbows flexed at 90°, with hands positioned 40 cm apart.
  The BlazePod unit will be placed centrally, approximately 20 cm away from each hand. When the BlazePod lights up, participants will be instructed to respond as quickly as possible by tapping the light to turn it off. As the lights will activate randomly, participants will be required to react unpredictably and respond accordingly each time the light appears.
  The total test duration will be recorded at the end of the trial.

OTHER OUTCOMES:
Fatigue Perception and Relief Sensation After Vibration or Rest | Change in baseline fatigue perception and relief sensation following intervention or rest
  To evaluate the effects of local vibration on fatigue perception and relief sensation, participants will be asked to rate the intensity of these two parameters on a scale from 0 to 10 before and after the application. A score of 0 indicates the lowest intensity, while a score of 10 represents an unbearable level.
Post-Fatigue Fatigue Rating | Change in baseline fatigue following muscle exhaustion protocol
  To evaluate the perception of fatigue emerging after the fatigue protocol, participants will be asked to rate the intensity of their fatigue on a scale from 0 to 10. A score of 0 indicates no fatigue, while a score of 10 represents an unbearable level of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: ömer dursun, Asst. Prof., Principal Investigator — Bitlis Eren University; merve tunçdemir, Asst. Prof., Principal Investigator — Bitlis Eren University
Locations (1):
- Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Bitlis Eren University, Bitlis, Turkey (Türkiye)

REFERENCES:
- [Background] Ferreira RM, Silva R, Vigario P, Martins PN, Casanova F, Fernandes RJ, Sampaio AR. The Effects of Massage Guns on Performance and Recovery: A Systematic Review. J Funct Morphol Kinesiol. 2023 Sep 18;8(3):138. doi: 10.3390/jfmk8030138. PMID 37754971
- [Background] Jones GC, Blotter JD, Smallwood CD, Eggett DL, Cochrane DJ, Feland JB. Effect of Resonant Frequency Vibration on Delayed Onset Muscle Soreness and Resulting Stiffness as Measured by Shear-Wave Elastography. Int J Environ Res Public Health. 2021 Jul 24;18(15):7853. doi: 10.3390/ijerph18157853. PMID 34360146
- [Background] Alam MM, Khan AA, Farooq M. Effects of vibratory massage therapy on grip strength, endurance time and forearm muscle performance. Work. 2021;68(3):619-632. doi: 10.3233/WOR-203397. PMID 33612507
- [Background] Chwala W, Pogwizd P, Rydzik L, Ambrozy T. Effect of Vibration Massage and Passive Rest on Recovery of Muscle Strength after Short-Term Exercise. Int J Environ Res Public Health. 2021 Nov 7;18(21):11680. doi: 10.3390/ijerph182111680. PMID 34770194
- [Background] Alam MM, Khan AA, Farooq M. Effect of whole-body vibration on neuromuscular performance: A literature review. Work. 2018;59(4):571-583. doi: 10.3233/WOR-182699. PMID 29733043
- [Background] Percival S, Sims DT, Stebbings GK. Local Vibration Therapy, Oxygen Resaturation Rate, and Muscle Strength After Exercise-Induced Muscle Damage. J Athl Train. 2022 May 1;57(5):502-509. doi: 10.4085/1062-6050-0064.21. PMID 35696601
- [Background] Liepert J, Binder C. Vibration-induced effects in stroke patients with spastic hemiparesis--a pilot study. Restor Neurol Neurosci. 2010;28(6):729-35. doi: 10.3233/RNN-2010-0541. PMID 21209488
- [Background] Kerschan-Schindl K, Grampp S, Henk C, Resch H, Preisinger E, Fialka-Moser V, Imhof H. Whole-body vibration exercise leads to alterations in muscle blood volume. Clin Physiol. 2001 May;21(3):377-82. doi: 10.1046/j.1365-2281.2001.00335.x. PMID 11380538
- [Background] Otadi K, Ghasemi M, Jalaie S, Bagheri H, Azizian M, Emamdoost S, Sarafraz H, Sepahvand M. A prophylactic effect of local vibration on quadriceps muscle fatigue in non-athletic males: a randomized controlled trial study. J Phys Ther Sci. 2019 Mar;31(3):223-226. doi: 10.1589/jpts.31.223. Epub 2019 Mar 19. PMID 30936635
- [Background] Ishikura H. Effects of local vibration stimulation on muscle recovery and hypertrophy. J Phys Ther Sci. 2024 Aug;36(8):441-446. doi: 10.1589/jpts.36.441. Epub 2024 Aug 1. PMID 39092417
- [Background] Rosenkranz K, Rothwell JC. Differential effect of muscle vibration on intracortical inhibitory circuits in humans. J Physiol. 2003 Sep 1;551(Pt 2):649-60. doi: 10.1113/jphysiol.2003.043752. Epub 2003 Jun 23. PMID 12821723
- [Background] Timon R, Tejero J, Brazo-Sayavera J, Crespo C, Olcina G. Effects of whole-body vibration after eccentric exercise on muscle soreness and muscle strength recovery. J Phys Ther Sci. 2016 Jun;28(6):1781-5. doi: 10.1589/jpts.28.1781. Epub 2016 Jun 28. PMID 27390415
- [Background] Fuller JT, Thomson RL, Howe PR, Buckley JD. Effect of vibration on muscle perfusion: a systematic review. Clin Physiol Funct Imaging. 2013 Jan;33(1):1-10. doi: 10.1111/j.1475-097X.2012.01161.x. Epub 2012 Aug 2. PMID 23216759
- [Background] Hogan MC, Richardson RS, Kurdak SS. Initial fall in skeletal muscle force development during ischemia is related to oxygen availability. J Appl Physiol (1985). 1994 Nov;77(5):2380-4. doi: 10.1152/jappl.1994.77.5.2380. PMID 7868458